CLINICAL TRIAL: NCT06565845
Title: Analysis of the Clinical Characteristics and Three Treatment Methods of Granulomatous Lobular Mastitis
Brief Title: Analysis of Various Treatment Methods of Granulomatous Lobular Mastitis
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024182
Record Dates: First submitted 2024-08-18; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Granulomatous Mastitis
Keywords: Granulomatous lobular mastitis; surgical treatment; antituberculosis therapy; surgery combined with anti-tuberculosis therapy
MeSH Terms: conditions — Granulomatous Mastitis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- surgery group: The patients underwent surgery
  Interventions: Procedure: Surgery
- triple anti-tuberculosis drug therapy group: The patients were treated with triple anti-tuberculosis drugs
  Interventions: Drug: triple anti-tuberculosis drug
- combination therapy group: The patients were treated with surgery first, and then took triple anti-tuberculosis drugs after surgery
  Interventions: Procedure: Surgery; Drug: triple anti-tuberculosis drug

INTERVENTIONS:
Procedure: Surgery — patients underwent complete excision of the inflammatory breast tissue and some surrounding normal tissue under combined intravenous with inhalation anesthesia. Damaged skin was also removed.
  Groups: combination therapy group; surgery group
Drug: triple anti-tuberculosis drug — Patients took oral rifampin (450 mg/day), isoniazid (300 mg/day), and ethambutol (15 mg/kg/day).
  Groups: combination therapy group; triple anti-tuberculosis drug therapy group

SUMMARY:
Granulomatous lobular mastitis (GLM) is a rare benign breast disease that is difficult to distinguish from breast cancer based on clinical and imaging findings, and there is currently no standard treatment. This study aims to analyze the clinical characteristics and demographic data of GLM patients and to compare the overall effectiveness of three treatment methods: surgery alone, triple anti-tuberculosis drug therapy alone, and combined surgery with triple anti-tuberculosis drug therapy, with the goal of providing new insights for clinical treatment.

DETAILED DESCRIPTION:
In recent years, the incidence of this disease has been increasing annually. The incidence of GLM is region-specific, being higher in Mediterranean regions and Asian countries. The etiology is currently unclear, but many studies suggest that GLM is associated with autoimmune disorders, hormonal imbalances, and microbial infections . GLM has a long course, is difficult to treat, and prone to recurrence, causing significant trauma to the patient's breast appearance and overall well-being. Currently, the main treatment methods for GLM include surgical treatment, drug therapy, combined surgery with drug therapy, and close observation. Surgical treatment options mainly include abscess incision and drainage, segmental resection, subcutaneous mastectomy, mastectomy, and breast reconstruction. Although surgical treatment can rapidly improve the condition, the recurrence rate reported in the literature ranges from 5% to 50% . Although GLM is a benign disease, it can severely impact the patient's normal life, causing physical and psychological trauma. However, few studies have included patients' subjective treatment experiences in the evaluation of treatment outcomes.

To date, there have been no studies comparing the efficacy of three treatment methods (surgery alone, triple anti-tuberculosis drug therapy alone, and combined surgery with triple anti-tuberculosis drug therapy) in the same population of GLM patients. This study aims to compare the efficacy and patient satisfaction of these three treatment methods, with the hope of providing new insights for clinical treatment options.

ELIGIBILITY:
Inclusion Criteria:

* non-lactating and aged 15-65 years
* histopathological confirmation of GLM
* normal liver and kidney function

Exclusion Criteria:

* lactating and pregnant women
* allergies to rifampin, isoniazid, or ethambutol
* concurrent malignant breast tumors
* severe underlying diseases
* other conditions deemed unsuitable by the investigator and
* refusal to participate in the study

Ages: 15 Years to 65 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Female patients with GLM who were treated at the Breast Surgery Department of the First Affiliated Hospital of Harbin Medical University were selected.Patients with GLM mostly present with unilateral disease, and the lesions can be located in any part of the breast. Arthritis and lower limb erythema nodosum are rare.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2024-09-19 (Estimated); Study Completion 2024-10-19 (Estimated)

PRIMARY OUTCOMES:
Differences in the cure rate of the three treatment modalities | Baseline
  According to the treatment method, the patients were divided into three groups: surgery group, triple anti-TB drug treatment group, and combination treatment group. IBM SPSS 27.0 software was used for statistical analysis. The cure rate was compared among the three groups.
Differences in the recurrence rate of the three treatment modalities | Baseline
  According to the treatment method, the patients were divided into three groups: surgery group, triple anti-TB drug treatment group, and combination treatment group. IBM SPSS 27.0 software was used for statistical analysis. The recurrence rate was compared among the three groups.
Differences in the incidence of adverse reactions of the three treatment modalities | Baseline
  According to the treatment method, the patients were divided into three groups: surgery group, triple anti-TB drug treatment group, and combination treatment group. IBM SPSS 27.0 software was used for statistical analysis. The incidence of adverse reactions was compared among the three groups.

SECONDARY OUTCOMES:
Differences in the patient satisfaction score (points) of the three treatment modalities | Baseline
  According to the treatment method, the patients were divided into three groups: surgery group, triple anti-TB drug treatment group, and combination treatment group. IBM SPSS 27.0 software was used for statistical analysis. The patient satisfaction score (points) was compared among the three groups.
Differences in the treatment duration (months) of the three treatment modalities | Baseline
  According to the treatment method, the patients were divided into three groups: surgery group, triple anti-TB drug treatment group, and combination treatment group. IBM SPSS 27.0 software was used for statistical analysis. The treatment duration (months) was compared among the three groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Feng, Study Director — First Affiliated Hospital of Harbin Medical University
Locations (1):
- First affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessler E, Wolloch Y. Granulomatous mastitis: a lesion clinically simulating carcinoma. Am J Clin Pathol. 1972 Dec;58(6):642-6. doi: 10.1093/ajcp/58.6.642. No abstract available. PMID 4674439
- [Background] Yuan QQ, Xiao SY, Farouk O, Du YT, Sheybani F, Tan QT, Akbulut S, Cetin K, Alikhassi A, Yaghan RJ, Durur-Subasi I, Altintoprak F, Eom TI, Alper F, Hasbahceci M, Martinez-Ramos D, Oztekin PS, Kwong A, Pluguez-Turull CW, Brownson KE, Chandanwale S, Habibi M, Lan LY, Zhou R, Zeng XT, Bai J, Bai JW, Chen QR, Chen X, Zha XM, Dai WJ, Dai ZJ, Feng QY, Gao QJ, Gao RF, Han BS, Hou JX, Hou W, Liao HY, Luo H, Liu ZR, Lu JH, Luo B, Ma XP, Qian J, Qin JY, Wei W, Wei G, Xu LY, Xue HC, Yang HW, Yang WG, Zhang CJ, Zhang F, Zhang GX, Zhang SK, Zhang SQ, Zhang YQ, Zhang YP, Zhang SC, Zhao DW, Zheng XM, Zheng LW, Xu GR, Zhou WB, Wu GS. Correction: Management of granulomatous lobular mastitis: an international multidisciplinary consensus (2021 edition). Mil Med Res. 2022 Aug 23;9(1):47. doi: 10.1186/s40779-022-00408-w. No abstract available. PMID 35999646
- [Background] Akcan A, Akyildiz H, Deneme MA, Akgun H, Aritas Y. Granulomatous lobular mastitis: a complex diagnostic and therapeutic problem. World J Surg. 2006 Aug;30(8):1403-9. doi: 10.1007/s00268-005-0476-0. PMID 16847715
- [Derived] Shang B, Zhang T, Liu C, Lu J, Cui C, Feng J, Zhou Y. Analysis of three treatment methods for granulomatous lobular mastitis: a retrospective study in a single center. Front Oncol. 2025 Apr 30;15:1588836. doi: 10.3389/fonc.2025.1588836. eCollection 2025. PMID 40371221